CLINICAL TRIAL: NCT05192993
Title: Effect of Oculomotor and Gaze Stability Exercise on Writing Capabilities on Autism
Brief Title: Effect of Oculomotor Exercise on Writing Capabilities on Autism
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Misr University for Science and Technology (Other)
Responsible Party: Principal Investigator, Samah Mahmoud Sheha, principal investigator, Misr University for Science and Technology
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/003283
Record Dates: First submitted 2021-10-21; First posted 2022-01-14 (Actual); Last update posted 2022-01-14 (Actual); Status verified 2021-12

CONDITIONS: Autism
MeSH Terms: conditions — Autistic Disorder

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- visual motor integration group (Experimental): participants in the experimental group will receive visual motor integration program
  Interventions: Other: visual motor integration group
- Handwriting intervention group (Active Comparator): participants in the experimental group will receive handwriting intervention program.
  Interventions: Other: Handwriting intervention programs
- visual motor integration and Handwriting intervention group (Active Comparator): participants in the group will receive visual motor integration program and handwriting intervention program.
  Interventions: Other: visual motor integration program and Handwriting intervention programs

INTERVENTIONS:
Other: visual motor integration group — Oculomotor exercises as follow:(1) Eye follow with a stationary head 2)Saccadic eye movements 3) Gaze stability 4)Eye/head co-ordination 5)Balancing exercises
  Arms: visual motor integration group
Other: Handwriting intervention programs — (1)Eye motor coordination (2)position in space(3)coping-figure ground(4)spatial relationship(5)visual closure(6)constancy of shapes(7)far and near coping
  Arms: Handwriting intervention group
Other: visual motor integration program and Handwriting intervention programs — Oculomotor exercises as follow:(1) Eye follow with a stationary head 2)Saccadic eye movements 3) Gaze stability 4)Eye/head co-ordination 5)Balancing exercises 6)Eye motor coordination (7)position in space(8)coping-figure ground(9)spatial relationship(10)visual closure(11)constancy of shapes(12)far and near coping
  Hand writing intervention as follow (1)Eye motor coordination (2)position in space(3)coping-figure ground(4)spatial relationship(5)visual closure(6)constancy of shapes(7)far and near coping
  Arms: visual motor integration and Handwriting intervention group

SUMMARY:
Autism spectrum disorders (ASD)are neurodevelopmental disorders that are clinically characterized by a triad of features: impairments in social interaction, impairments in communication, and presence of restrictive repetitive and stereotypical behaviors, interests, or activities (DSM-IV). In addition to these core deficits, ASD is associated with a high prevalence of fine motor difficulties and executive function impairments that contribute to acquisition and performance of skilled motor tasks. It is therefore not surprising that handwriting difficulties are frequently reported in children with ASD.

DETAILED DESCRIPTION:
Handwriting is a functional skill that profoundly affects children's academic and psychosocial development. Difficulties in acquiring and applying these skills subsequently lead to problems such as slow writing and illegible written .Such difficulties may have implications on the child's successful participation in school and play activities, potentially leading to problems in academic performance and lowered self-esteem .Therefore, students with handwriting difficulties are especially prone to frustration, disappointment, and under achievement. The aim of our study is to improve handwriting quality of children with ASD.

ELIGIBILITY:
Inclusion Criteria:

* Mild autism (score 55-71) on Gilliam Autism Rating Scale (GARS-3).
* Intelligence quotient (IQ) score 70-100.
* Writing difficulties

Exclusion Criteria:

* Middle ear disorders
* Physical or mental conditions that may affect handwriting (e.g., seizures)
* Uncorrected visual or hearing impairments.

Ages: 5 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-03 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
gaze stability | 6 weeks
  Rating scale of gaze stability
  0= negative Gaze stable smooth well coordinated,percise and fast movement of the head,fluent change of head movement direction
  1. modreate positive Gaze stable,slightely irregular head movement
  2. strong positive Gaze repeatedly unstable ,head movement slow and irregular

SECONDARY OUTCOMES:
eye head coordination | 6 weeks
  Rating scale of sequential head and eye movements 0= negative Clear,regular ,smooth, dissociated movements,of head and eyes.
  1. moderately positive slightely decelerated eye movements.occasional associated eye-head movements ,head unstable.
  2. strongly positive clearly decelerated , irregular and often associated eye -head movements test not feasible.

OTHER OUTCOMES:
saccadic eye movement | 6 weeks
  0= negative Smooth, percise, fast eye movements,fast change of gaze direction,head remain stable
  1. moderately positive slightely irregular eye movements.Short stops before changing gaze direction.Head slightly unstable
  2. strongly positive Eye movements clearly slower or irregular.Prolonged maintenance of gaze direction before changing direction.Obvious head movement.Test cannot be performed.

CONTACTS AND LOCATIONS:
Overall Officials: Samah M Sheha, PhD, Principal Investigator — Misr University for Science and Technology
Locations (1):
- Misr university for science and technology, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Accardo AL, Finnegan EG, Kuder SJ, Bomgardner EM. Writing Interventions for Individuals with Autism Spectrum Disorder: A Research Synthesis. J Autism Dev Disord. 2020 Jun;50(6):1988-2006. doi: 10.1007/s10803-019-03955-9. PMID 30838491